CLINICAL TRIAL: NCT01557569
Title: Clinical Efficacy of Atomoxetine for Methamphetamine Dependence
Acronym: ATM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 133414
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Methamphetamine Dependence
Keywords: methamphetamine; addiction; relapse; atomoxetine
MeSH Terms: conditions — Behavior, Addictive; Recurrence | interventions — Atomoxetine Hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atomoxetine (Active Comparator): Group receiving atomoxetine
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): Group will receive placebo instead of atomoxetine
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Atomoxetine — During the first 2 weeks and three days the dose of atomoxetine will be titrated up starting with 20 mg/day for first 3 days, 36 mg/day for next 4 days, 50 mg/day for next 3 days, and finally 80 mg/day until the final day of the study (week 10, day 7)
  Other Names: strattera
  Arms: Atomoxetine
Drug: placebo — participants in this group will receive 1 dose of placebo daily for the entire 10-weeks.
  Other Names: "sugar pill"
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the ability of atomoxetine compared to placebo to increase time to relapse in methamphetamine dependent volunteers. Our hypothesis is that atomoxetine will increase time before (if) the participant relapses.

DETAILED DESCRIPTION:
During the study participants will spend the initial 2-weeks of the study at an inpatient facility. This will help participants initiate withdrawal. During the following 8-weeks the participant will come in for 3-4 visits each week. Three of these visits will be with the research assistants and one visit will be with a therapist in order to work with the participant using a cognitive behavioral therapy approach. Therapy visits are typically scheduled on a day that the participant is coming for clinic anyways so the number of visits per week is typically 3. During the 10-week period the investigators will collect various measures, including vitals, cognitive assessments, mood assessments, urine drug screens, weekly use reports of methamphetamine, and any reports of symptoms or side effects. This will tell the investigators if atomoxetine is safe and if a participant lapsed or relapsed.

ELIGIBILITY:
Inclusion Criteria.

* 18-65 years old
* Seeking treatment for METH use
* METH dependence, as assessed by the substance abuse section of the Structured Clinical Interview for DSM-IV.
* At least weekly self-reported METH use during a preceding three month period
* Women of childbearing age must have a negative pregnancy test, agree to adequate contraception to prevent pregnancy during the study, agree to monthly pregnancy testing, and not be nursing
* Men must agree to use effective means of contraception during the study.

Exclusion Criteria.

* Suicide attempts within the past 12 months or either suicidal ideations or psychotic symptoms in the past 6 months as determined by a study physician.
* Current opioid, alcohol or sedative physical dependence or cocaine dependence
* Major cardiovascular disorder that contraindicates study participation (e.g., history of myocardial infarction, stroke, congestive heart failure, cardiac arrhythmia, hypertension [i.e., > 160 SBP or > 100 DBP] or an unstable medical condition (e.g., untreated bacterial infection) as determined by the study physician.
* Schizophrenia or bipolar disorder of any type
* Present or recent use (within 2 weeks) of over-the-counter or prescription drug that would be expected to have major interaction with atomoxetine (e.g., an monoamine oxidase inhibitor (MAOI), paroxetine, fluoxetine, quinidine, dopamine, albuterol, or other β2-agonists)
* Medical contraindication to receiving atomoxetine (e.g., severe hepatic impairment, glaucoma, heart disease, hypertension, seizure disorders, documented hypersensitivity to atomoxetine); or other bronchospastic condition, (2nd or 3rd degree AV block, sick sinus rhythm, severe hepatic impairment, documented hypersensitivity to atomoxetine)
* Liver function tests (i.e., liver enzymes) greater than two times normal levels
* Systolic blood pressure of < 90 or > 160 mmHg, diastolic blood pressure of < 60 or > 100 mmHg, or sitting heart rate of < 55 or > 100 beats/min or blood pressure readings > 140 systolic or > 90 diastolic on three separate, consecutive occasions.
* History of pheochromocytoma
* Pregnant or nursing female

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Oliveto, PhD, Principal Investigator — University of Arkansas
Locations (1):
- UAMS, Psychiatric Research Institute, Center for Addiction Research, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atomoxetine | Placebo
Started | 6 (Those who received at least one dose of medication) | 7 (Those who received at least one dose of medication)
Completed 2-wk Residential Stay | 3 | 1
Completed | 1 | 0
Not Completed | 5 | 7
Not completed — Adverse Event | 2 | 0
Not completed — high blood pressure | 0 | 1
Not completed — Withdrawal by Subject | 3 | 5
Not completed — noncompliance with rules of residential | 0 | 1

BASELINE CHARACTERISTICS:
Population: those that received at least one dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Time Till Relapse
Description: The number of days until a participant has a relapse, which will be measured by qualitative urine drug screens. To ensure a large enough sample, those who drop out prior to completing the residential stay will be included in this analysis (with minus days until relapse)
Time Frame: 57 days
Population: Only 4 of 13 finished the 2-week residential stay. Since subjects who drop out are deemed relapsed, all subjects receiving >/=1 dose of study med were included in the analyses. Those who dropped out before completing the residential stay were considered relapsed by the second day and the date of discharge was subtracted from this relapse date.
Measure: Median (Full Range); unit: Days to Relapse
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 6 | 7
Days to Relapse | 7 [-10 to 57] | -8 [-12 to 27]
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Due to skewed data, Kruskal Wallis Test was used; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis; Median Difference (Final Values) = 0.413

ADVERSE EVENTS:
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 4/6 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=6) | Placebo (N=7)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
sharp apin/tingling in limb (Nervous system disorders) | 1 (1) | 0 (0)
sleepiness/tiredness (General disorders) | 1 (1) | 1 (1)
night sweats (General disorders) | 1 (1) | 0 (0)
elevated BP (outside parameters) (Cardiac disorders) | 0 (0) | 1 (1)
elevated BP on 3 separate occasions (Cardiac disorders) | 0 (0) | 1 (2)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
insomnia (General disorders) | 2 (2) | 0 (0)
rapid heartbeat (Cardiac disorders) | 2 (3) | 0 (0)
irritability (Psychiatric disorders) | 1 (1) | 0 (0)
dry mouth (General disorders) | 1 (1) | 0 (0)
hot flash (General disorders) | 1 (1) | 0 (0)
chest pain (Cardiac disorders) | 1 (1) | 0 (0)
labored breathing (General disorders) | 1 (1) | 0 (0)
headache/pain (Nervous system disorders) | 1 (2) | 0 (0)
nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment and retention was much more difficult than anticipated. Because of, this too few (3 in ATM and 1 in PLA) were retained through the residential stay to determine efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes